CLINICAL TRIAL: NCT02751008
Title: Bone Fragility Study in Pediatric Population With Risk Factors
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FRA-2016-11
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Bone Loss, Age-Related
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Low bone mass and osteoporosis are underdiagnosed in childhood in our environment and its prevalence is unknown. In most cases they are secondary to chronic diseases that conduct to a poor bone health condition and thereby a risk of fracture increased. The aim of this study is to identify patients with risk factors for low bone mass and determine their Bone Mineral Density (amount of bone) by performing bone densitometry and compared with healthy population of the same characteristics. Also the investigators want to evaluate bone quality by application of Trabecular Bone Score to images obtained by densitometry. As secondary objectives the investigators intend to correlate the data with with clinical variables to identify the most important in bone health clinical factors. In addition to measuring bone quality and quantity demographic and clinical process related to bone quality base and variables will be collected.

DETAILED DESCRIPTION:
Osteoporosis (OP) in children is a rare disease whose incidence is unknown, partly due to lack of diagnosis associated with the absence of specific clinical symptoms in the early stages of the disease.

That is why the active recognition of this disease by the pediatrician and the pediatrician rheumatologist is essential to prevent future complications: fractures and comorbidity associated with them, including possible deformities and the need for surgical correction.

The diagnosis of OP in children and adolescents requires the combination of densitometric criteria (low bone mass or deficits in mineralization) and the clinical judgment of clinically significant fracture. Any of the following fractures are considered clinically significant fractures: Long bone fracture of the lower limbs, vertebral compression fracture, or two or more long bone fractures of upper extremities.

Low bone mass for age is considered when the Z-score of the measurement of bone mineral density (BMD) is less than or equal to -2, adjusted for age, sex and body mass index.

The Z-score is a value that is calculated by subtracting the average patient BMD BMD their age group and gender and this value by dividing the standard deviation of their age group and gender.

DXA (dual-energy X ray absortiometry) lumbar and whole body (excluding the head) is the method of choice for measuring bone mineral density (BMD), since it is the most accurate skeletal location and reproducible for measuring BMD.

Juvenile Idiopathic Osteoporosis is a very rare entity, with less than 200 cases described in the literature, and whose diagnosis requires the exclusion of secondary forms of osteoporosis.

Among the causes of osteoporosis (low bone mass or) secondary in child population the investigators have: kidney diseases, metabolic diseases, hematological, endocrinological, gastrointestinal and rheumatological, including chronic systemic disorders. The transplant and cancer patients have generally a multifactorial risk of osteoporosis (immobilization, medical treatment, etc.).

Also, nutritional causes are another large block of secondary forms of child and / juvenile (or low bone mass for age) osteoporosis. Typical examples of malabsorptive disease are celiac disease, cystic fibrosis and chronic inflammatory bowel disease and anorexia nervosa.

Special attention should pediatric patients treated with nonsteroidal antiinflammatory drugs, methotrexate and, of course, glucocorticoids, potent inducers and inhibitors of osteoclastogenesis osteoblastogenesis.

Other medications that affect a greater risk of developing osteoporosis are: some anticonvulsants, anticoagulants and chemotherapies.

According to the ISCD (International Society for Clinical Densitometry) should be performed by DXA bone densitometry as a measure of bone health assessment of all children with increased risk of fracture. They are therefore candidates for a bone densitometry pediatric patients with primary bone diseases or potential secondary bone diseases (eg, pre-transplant chronic inflammatory diseases, endocrine disorders, cancer or history).

While DXA is the only validated technique today for indirect measurement of fracture risk in itself is only able to analyze changes in bone mineral content, so recently they have intensified efforts to validate other techniques possible to assess not only the quantity but also the quality of the bone. Among the highlights is the TBS (Trabecular Bone Score) which is software that applied directly to the information obtained through the spinal DXA can analyze the trabecular number, thickness and connectivity, providing extra information about the strength or weakness of the vertebra. Its use is spreading in routine clinical practice in the adult population as it is safe and does not increase the time required exploration, however in the pediatric population is not included in routine practice even though its application could provide additional information to the DMO on which to base treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 21 years of age who are at risk of bone fragility ( according to criteria previously set forth in the background section ) and whose parents / guardians have signed the informed consent

Exclusion Criteria:

* Subjects who refuse to participate in the study. Over 16 years old. Bone prior active treatment .

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients under 21 years of age who are at risk of bone fragility (pediatric patients with primary bone diseases or potential secondary bone diseases (eg , chronic inflammatory diseases , endocrine disorders , history of cancer or pre- transplant) and whose parents / guardians have signed the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Bone mass | 1 day visit

SECONDARY OUTCOMES:
Bone quality | 1 day visit
  Performing Trabecular Bone Score vapplied directly to the information obtained through the spinal DXA

IPD SHARING:
Plan to Share IPD: Undecided